CLINICAL TRIAL: NCT00396110
Title: Evaluation of the Efficacy of Rosuvastatin in Daily Practice (TARGET)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: 25V06; TARGET
Record Dates: First submitted 2006-11-03; First posted 2006-11-06 (Estimated); Last update posted 2006-11-06 (Estimated); Status verified 2003-02

CONDITIONS: Hypercholesterolemia; Coronary Heart Disease
Keywords: cholesterol; coronary heart disease; rosuvastatin; LDL-C goal; hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
In this study the effect of the switch to rosuvastatin from another statin (fluvastatin, pravastatin, simvastatin, atorvastatin) was evaluated in high-risk patients with and without evident CHD and LDL-C ≥ 3.2 mmol/l. This was done in a large observational study (TARGET) representing daily practice. Primary end points analysis was the percentage of patients reaching the target of LDL-C < 3.2 mmol/l. Secondary outcomes were the changes of LDL-C, HDL-C, TC, Triglycerides (TG) and TC/HDL-C-ratio from baseline.

ELIGIBILITY:
Inclusion Criteria:

* High-risk patients with and without evident CHD who had LDL-C > 3.2 mmol/l and were treated at that moment with HMG-CoA-reductase inhibitor apart from rosuvastatin.
* Patients were aged >18 years and <70 years (men) and < 75 years (women).

Exclusion Criteria:

* Treatment with atorvastatin 40 or 80 mg or simvastatin 80 mg
* Patients familiar with muscular pain, myopathy or liver function disorders (inclusive elevation of serum transaminases) and/or contra-indications for treatment with rosuvastatin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3889
Dates: Start 2003-02

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid van Geel, MD, Study Chair — AstraZeneca; Ingeborg Vosjan, MD, Study Chair — AstraZeneca